CLINICAL TRIAL: NCT06108271
Title: Innovative Endotracheal Tube Design Reduces Postoperative Laryngeal Injury
Acronym: Triglotix®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of the Nuestra Señora de Candelaria (Other)
Responsible Party: Principal Investigator, Pedro Luis Bravo, Director, University Hospital of the Nuestra Señora de Candelaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Endotracheal tube Triglotix®
Record Dates: First submitted 2023-09-27; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Laryngeal Injury; Hoarseness; Cough; Sore-throat; Intubation Complication; Bucking, Anesthesia Related
Keywords: Laryngeal Injury; Endotracheal tube; General anesthesia
MeSH Terms: conditions — Hoarseness; Cough; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETT-T (Experimental): Endotracheal tube Triglotix®
  Interventions: Device: Triglotix®
- ETT-C (Active Comparator): Endotracheal tube conventional
  Interventions: Device: Conventional endotracheal tube

INTERVENTIONS:
Device: Triglotix® — The Triglotix® has a biocompatible self-expanding viscoelastic cuff that is located in the supraglottic, glottic and subglottic space. This cuff separates the endotracheal tube from the laryngeal vestibule in the supraglottic space and the vocal cords avoiding direct tissue damage from the plastic components of the tube. The viscoelastic cuff self-expands after the endotracheal tube is in adequate position in the airway. Then it adapts progressively and gradually to the shape of structures it comes in contact with, applying minimal pressure to the surrounding tissue. The ETT-T also has two wire reinforced segments: the first is located outside the mouth to prevent deformation related with kinking, while the second segment is positioned distally along the larynx. The primary purpose of this design is to mitigate torsional, rotational and lateralization forces that the tube may encounter while the patient is intubated.
  Other Names: ETT-T
  Arms: ETT-T
Device: Conventional endotracheal tube — Conventional endotracheal tube that is currently used worldwide
  Other Names: ETT-C
  Arms: ETT-C

SUMMARY:
The goal of this randomized clinical trial is to compare two different orotracheal tubes in patients which require orotracheal intubation for general anesthesia. The main questions it aims to answer are:

* To assess the presence of laryngeal injury
* To evaluate the consequences in voice quality
* To ask for the presence of symptoms as sore throat, hoarseness, and cough

Participants will be randomly assigned into two groups, one will use conventional endotracheal tube and the other will use Triglotix® endotracheal tube.

DETAILED DESCRIPTION:
Endotracheal intubation is necessary in some patients undergoing surgical procedures and patients requiring mechanical ventilation in the intensive care unit. However, endotracheal intubation is associated with known complications. In post-surgical patients subjected to orotracheal intubation, the incidence of dysphagia, sore throat, hoarseness and cough is 43%,38%27%,32% respectivelly. These figures increase in cases of prolonged intubation, such as those in intensive care units, where reported rates are 76% for sore throat, 63% for hoarseness and 49% for dysphagia. No significant endotracheal tube design improvements have been developed over the past few decades addressing these issues.

The present study aims to compare the incidence of laryngeal injuries, and related symptoms as sore throat, hoarseness, swallowing problems, bucking and coughing between two defined sample populations: those utilizing a conventional endotracheal tube (ETT-C) and those employing the new Triglotix® endotracheal tube (ETT-T) in patients undergoing elective surgery requiring general anesthesia and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Elective perianal surgery requiring intubation for general anesthesia
* Duration range 30-90 minutes

Exclusion Criteria:

* Difficult airway
* American Society of Anesthesiologists physical status (ASA) > III
* Morbid obesity (body mass index >40 kg/m2)
* Patients not suitable for outpatient surgery
* Patients with history of previous neck surgery
* Patients with history of dysphagia
* Patients with comorbidities as diabetes and hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Laryngeal injury | Immediately before the induction and 45 minutes after the end of the procedure
  Laryngeal pathology was assessed based on the location (unilateral: right/left or bilateral) and on morphology: grade 0 = no lesions, grade 1 = superficial erythema (redness of the mucosa without surrounding inflammation), grade 2 = oedema (swollen mucosa at the vocal cords), grade 3 haematoma (redness of the mucosa with surrounding inflammatory swelling), grade 4 = mucosal laceration (causing active bleeding into the vocal cords), grade 5 = arytenoid dislocation or subluxation (arytenoid with limited movement), and grade 6 = vocal cord palsy

SECONDARY OUTCOMES:
Postoperative cough | 45 minutes after the end of the procedure
  Postoperative cough was assessed: (0 = None, 1 = mild cough, 2 = moderate cough <5 s, 3 = Severe cough >5 s)
Bucking during extubation | During extubation
  Presence of bucking during extubation assessed by the anesthesiologist just after stimulating the patient (1 = mild, 2 = severe, 3 = abscense)
Acoustic Voice Quality Index 03.01 (AVQIv3) | Immediately before the induction and 45 minutes after the end of the procedure
  Concatenated voice samples of 3 seconds of sv [a:] and voiced segments of a phonetically balanced text.
Acoustic Breathiness Index (ABI) | Immediately before the induction and 45 minutes after the end of the procedure
  Concatenated voice samples of 3 seconds of sv [a:] and voiced segments of a phonetically balanced text.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Bravo, MD, Principal Investigator — University Hospital of the Nuestra Señora de Candelaria
Locations (1):
- Pedro Luis Bravo, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available six months after the end of the analysis.
Access Criteria: Main investigator is the contact for review requests

REFERENCES:
- [Background] Mendels EJ, Brunings JW, Hamaekers AE, Stokroos RJ, Kremer B, Baijens LW. Adverse laryngeal effects following short-term general anesthesia: a systematic review. Arch Otolaryngol Head Neck Surg. 2012 Mar;138(3):257-64. doi: 10.1001/archoto.2011.1427. PMID 22431870
- [Background] Melsen WG, Rovers MM, Groenwold RH, Bergmans DC, Camus C, Bauer TT, Hanisch EW, Klarin B, Koeman M, Krueger WA, Lacherade JC, Lorente L, Memish ZA, Morrow LE, Nardi G, van Nieuwenhoven CA, O'Keefe GE, Nakos G, Scannapieco FA, Seguin P, Staudinger T, Topeli A, Ferrer M, Bonten MJ. Attributable mortality of ventilator-associated pneumonia: a meta-analysis of individual patient data from randomised prevention studies. Lancet Infect Dis. 2013 Aug;13(8):665-71. doi: 10.1016/S1473-3099(13)70081-1. Epub 2013 Apr 25. PMID 23622939
- [Background] Brodsky MB, Akst LM, Jedlanek E, Pandian V, Blackford B, Price C, Cole G, Mendez-Tellez PA, Hillel AT, Best SR, Levy MJ. Laryngeal Injury and Upper Airway Symptoms After Endotracheal Intubation During Surgery: A Systematic Review and Meta-analysis. Anesth Analg. 2021 Apr 1;132(4):1023-1032. doi: 10.1213/ANE.0000000000005276. PMID 33196479
- [Background] Brodsky MB, Levy MJ, Jedlanek E, Pandian V, Blackford B, Price C, Cole G, Hillel AT, Best SR, Akst LM. Laryngeal Injury and Upper Airway Symptoms After Oral Endotracheal Intubation With Mechanical Ventilation During Critical Care: A Systematic Review. Crit Care Med. 2018 Dec;46(12):2010-2017. doi: 10.1097/CCM.0000000000003368. PMID 30096101
- [Background] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Background] Delgado Hernandez J, Leon Gomez NM, Jimenez A, Izquierdo LM, Barsties V Latoszek B. Validation of the Acoustic Voice Quality Index Version 03.01 and the Acoustic Breathiness Index in the Spanish language. Ann Otol Rhinol Laryngol. 2018 May;127(5):317-326. doi: 10.1177/0003489418761096. Epub 2018 Feb 28. PMID 29490478
- [Background] Mencke T, Echternach M, Kleinschmidt S, Lux P, Barth V, Plinkert PK, Fuchs-Buder T. Laryngeal morbidity and quality of tracheal intubation: a randomized controlled trial. Anesthesiology. 2003 May;98(5):1049-56. doi: 10.1097/00000542-200305000-00005. PMID 12717124
- [Background] Bishop MJ. Mechanisms of laryngotracheal injury following prolonged tracheal intubation. Chest. 1989 Jul;96(1):185-6. doi: 10.1378/chest.96.1.185. No abstract available. PMID 2661158
- [Background] Weymuller EA Jr, Bishop MJ, Fink BR, Hibbard AW, Spelman FA. Quantification of intralaryngeal pressure exerted by endotracheal tubes. Ann Otol Rhinol Laryngol. 1983 Sep-Oct;92(5 Pt 1):444-7. doi: 10.1177/000348948309200506. PMID 6625441
- [Result] Sajedi P, Maaroffi V. The macroscopic changes of tracheal mucosa following tight versus loose control of tracheal tube cuff pressure. Acta Anaesthesiol Sin. 2002 Sep;40(3):117-20. PMID 12434607
- [Derived] Bravo PL, Gonzalez Sammarco F, Cueva Nieves DA, Lorente L, Delgado J, Martinez-Ruiz R. Innovative Endotracheal Tube Design Reduces Laryngeal Injury with an Excellent Airway Seal and Minimal Cuff Pressures. Anesth Analg. 2025 Apr 1;140(4):983-985. doi: 10.1213/ANE.0000000000007260. Epub 2024 Oct 17. No abstract available. PMID 39418198